CLINICAL TRIAL: NCT05518344
Title: Clinical Investigation of "Viziatek ISL™ Refractive Phakic Intra Sulcus Lens" for Refraction Adjustment in Blind Volunteers
Brief Title: Study of Viziatek ISL™ Refractive Phakic Intra Sulcus Lens for Refraction Adjustment in Blind Volunteers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision to terminate the study
Sponsor: Hanita Lenses (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VZT-19-002
Record Dates: First submitted 2021-03-09; First posted 2022-08-26 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Experimental): * Release ISL from Inserter
  * Remove Inserter.
  * Tack the haptics under the iris in 4 locations
  * Verify that ISL is centered
  * Remove lid speculum and drape from subject's eye and face.
  * Move the subject to a slit lamp and verify ISL centration.
  Interventions: Device: Viziatek ISL™ (hereinafter referred to as the "ISL") implanted in blind eye.

INTERVENTIONS:
Device: Viziatek ISL™ (hereinafter referred to as the "ISL") implanted in blind eye. — Viziatek ISL™ (hereinafter referred to as the "ISL") implanted in blind eye.

SUMMARY:
This is a clinical investigation. A total of up to 5 subjects, but not less than 3 at one investigational site will undergo insertion of the ISL in one eye and will be followed through 6 months postoperative.

Subjects from the United States will not be enrolled in this study.

DETAILED DESCRIPTION:
The Viziatek ISL is intended to improve myopic vision and decrease dependence on glasses in myopic adults who don't have an irregular astigmatic cornea (as evaluated by topography), who require correction of -3.50 D to -23 D, who have BCVA - Distance between 20/20 to 20/30 and with no more than 5 D of the refractive cylinder, and who have stable MRSE within 0.50 D over the past 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must sign and be given a copy of the signed Informed Consent Form (ICF).
2. Subjects must be legally blind.
3. Subjects must have best-corrected distance visual acuity of 20/400 or worse.
4. Subjects must have an endothelial cell count ≥ 1800 cells/mm2 in the eye to be implanted.
5. Subjects must have a photopic pupil size of > 2 mm in the eye to be implanted.
6. Anterior chamber depth (ACD) ≥ 2.8 mm
7. Anterior chamber angle ≥ Grade III
8. Subjects must be willing and able to return for scheduled follow-up examinations for 12 months after surgery if asked.

Exclusion Criteria:

1. Subjects who have best-corrected visual acuity of better than 20/400
2. Subjects with clinically significant anterior segment pathology, including cataracts, in either eye.
3. Subjects with residual, recurrent, active ocular or uncontrolled eyelid disease or any progressive corneal abnormalities (including endothelial dystrophy, guttate in the central cornea, etc.) in the eye to be treated.
4. Subjects with a history of the chronic dry eye not controlled on therapy or with superficial punctuate keratitis (SPK) grade > II (i.e., greater than mild) based on Oxford Grading Scale12 in the eye to be treated.
5. Subjects who have undergone previous intraocular or corneal surgery including cataract and refractive surgery (e.g., LASIK surgery) in either eye.
6. Subjects using ophthalmic medication(s) other than artificial tears for treatment of ocular pathology.
7. Subjects with a history of autoimmune disease, connective tissue disease, or clinically significant atopic syndrome.
8. Subjects with a history of herpes zoster or herpes simplex keratitis.
9. Subjects with a history of a steroid-responsive rise in intraocular pressure (IOP), or a preoperative IOP > 21 mmHg or glaucoma.
10. Subjects with distorted, non-reactive, or decentered pupils.
11. Subjects on chronic systemic or topical corticosteroids or other immunosuppressive therapy that may affect wound healing, and any immuno-compromised subjects (use of intranasal steroids for seasonal allergies are acceptable).
12. Subjects using systemic medications with significant ocular side effects.
13. Subjects who are pregnant or are considering becoming pregnant during the time of the study.
14. Subjects with known sensitivity to planned study concomitant medications.
15. Subjects who are participating in any other drug or device clinical investigation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-06-04 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-03-16 (Actual)

PRIMARY OUTCOMES:
Endothelial cell loss | 6 months
  Endothelial cell loss in operated eye measured at months 6, and change in cell count from baseline less than 10%.

SECONDARY OUTCOMES:
Ultrasound Biomicroscopy (UBM) | 6 months
  All patients will undergo measurement of the central distance between implanted lens and anterior capsule to be greater than 50 microns (µm)

OTHER OUTCOMES:
Slit Lamp Examination | 6 months
  This includes measurement of aqueous cell and flare by a standard grading system and an evaluation for presence of corneal abnormalities; pupillary irregularities; iris atrophy and pigment dispersion
Pupillometry | 6 months
  Pupil diameter in bright light (photopic condition): 2-4 mm Pupil diameter in the dark (mesopic/scotopic conditions): 4-8 mm The pupils are generally equal in size. Pupil diameter is measured by digital pupilometer that measures distance between the center of each pupil.
Keratometry | 6 months
  Measurement of the power of the cornea
Best corrected Visual Acuity | 6 months
  Measurement by looking at ETDRS Chart with glasses

CONTACTS AND LOCATIONS:
Locations (1):
- Drsolomatinisilmakeskus, Riga, Latvia